CLINICAL TRIAL: NCT02592005
Title: Impact of Particulate Matter on Mothers and Babies in Antwerp (IPANEMA), a Prospective Cohort Study on the Impact of Pollutants and Particulate Matter in Pregnancy: Methodology and Design
Brief Title: Impact of Particulate Matter on Mothers and Babies in Antwerp (IPANEMA)
Acronym: IPANEMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Prof Yves Jacquemyn, Head of Obgyn, Universiteit Antwerpen
Other Study IDs: 14/40/411
Record Dates: First submitted 2015-10-22; First posted 2015-10-30 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Pregnancy; Preeclampsia
Keywords: pollution
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — maternal blood maternal hair maternal urine umbilical cord blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: amount of fine dust and other environmental exposure — this study compares levels of exposure to to fine dust PM 2.5 by individual measurement both at home and at work

SUMMARY:
Introduction: An emerging body of evidence indicates that there is an association between air pollution exposure in pregnancy and adverse pregnancy outcomes (Rudra, Williams, Sheppard , Koenig, & Schiff, 2011; Dadvand, et al., 2013; Ritz, et al., 2014). Adverse pregnancy outcomes tend to lead to adverse neonatal outcome and a higher economic cost. Epidemiologic studies have also revealed that cardiovascular complications during pregnancy, such als preeclampsia, are associated with a greater cardiovascular risk during later life ( Abramson & Melvin, 2014).

Aim: This study wants to examine the effects of exposure to environmental factors, polluents and particulate matter on the clinical pregnancy outcome for mother and child and to determine which biochemical changes in maternal, placental and cord blood best explain this effect.

Methods: This study will be performed in a prospective cohort setup (n=200), recruited from the prenatal clinic in the University Hospital Antwerp. The data collection consists of four questionnaires (intake, both urine samples and postpartum), two blood samples (28 weeks and post-partum), two urine samples (20 and 30 weeks), two hair samples (20 weeks and post-partum), cord blood and the placenta.

Results and conclusion: As the study will start in November 2014, no results are available yet.

DETAILED DESCRIPTION:
Blood collections (maternal and umbilical cord) Venous blood is drawn around 24 weeks of gestational age.

Table 1 Tests on maternal blood sample:Routine blood sampling (UZA) Urea, Creatinin, CRP, LDH, AST, ALT, Uric acid, APTT, PT, Fibrinogen, D-dimers, Glucose, Erythrocytes/hematocrit, Hemoglobin, Thrombocytes, Leukocytes, Ferritin, Toxoplasmosis (IgG & IgM), CMV (IgG & IgM), Herpes simplex IgG, Varicella zoster IgG, Rubella IgG, Parvovirus (IgG & IgM), Syphilis (RPR & TPHAM), Indirect Coombs AML sFlt-1, PlGF, Cystatin C VITO m(i)RNA expression, telomere length, DNA methylation

Umbilical cord blood is taken at time of birth. Table 2 Tests on umbilical blood sample VITO m(i)RNA expression, telomere length, DNA methylation

Urine collections Urine samples are taken by the pregnant women themselves, after a minimum of 8 hours fasting (morning urine). Samples are handed to the midwife at the antenatal visit, and placed at -20°C freezer within 12 hours of collection. Analysis will be performed at the Flemish Institute for Technological Research (VITO).

Two urine samples are collected: at 20 weeks and at 30 weeks gestational age. 8 oxo deoxyguanosine will be determined in the samples.

Hair collections Hair samples are drawn by the midwife around 24 weeks of gestational age and three days after delivery. Long periods of stress are associated with increased hair cortisol concentrations (Stalder & Kirschbaum, 2012). Confounding variables are low maternal education, season of delivery, smoking during pregnancy and obesity (Braig, et al., 2015).Titanium scissors are cleaned with denaturated ethanol and the midwife wears disposable gloves in order to limit contamination. A lock of hair with a thickness of a match (2 mm) and a length of 4 cm will be taken and put in an envelope. Analysis will be performed at the University of Southern Denmark.

Collection of particulate matter on bedroom window Participants will be asked to clean their bedroom window with clear water on the in- and outside around 24 weeks of gestation. A poster (A4 format) will then be attached to the window to create a standardized area for the measurement of magnetic particles. After minimal 4 weeks, the area in the poster is cleaned with a sterile pre-injection swab, on both sides of the window. Swabs are transported in a plastic bag and the ferro(i)magnetic particulate matter fraction will be quantified by Saturated Isothermal Remanent Magnetization.

Questionnaires

There are four different questionnaires:

Questionnaire on general habits, socio-economic factors, lifestyle and eating habits A self-designed questionnaire is used to extensively collect information on ethnic origin and and education level, on employment, income and work environment, on family history of diseases and chronic disorders, on eating habits, on previous pregnancies and other habits (smoking, alcohol consumption).

Questionnaire on lifestyle during previous 3 days A self-designed questionnaire is used to extensively collect information on contact with possible toxic factors and on eating pattern of the previous 3 days.

Questionnaire on residential facts A self-designed questionnaire is used to collect information about the exact location of the bedroom window and other possible factors influencing concentrations of particulate matter.

Questionnaire on stress factors and birth facts A self-designed questionnaire is used to extensively collect information on stress levels during pregnancy, on birth facts and on medication during pregnancy.

Questionnaires will be taken at different visits:< 12 weeks 20 weeks 30 weeks birth Questionnaire on general habits, socio-economic factors, lifestyle and eating habits Recruitment Questionnaire on lifestyle during previous 3 days Urine sample 1 Urine sample 2 Questionnaire on residential facts 4-8 weeks prior to visit Questionnaire on stress factors and birth facts 3 days after birth

ELIGIBILITY:
Inclusion Criteria:

* A singleton pregnancy from 12 weeks of gestational age
* Delivery planned in a hospital within the network of the Antwerp University
* Dutch speaking

Exclusion Criteria:

* Multiple pregnancy
* Planned home delivery of in another hospital

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women are recruited within the network of the Antwerp University. Leading centre will be the University Hospital Antwerp (UZA),a tertiary centre with a maternal intensive care unit (MIC) and a neonatal intensive care unit (NIC) and 1000 deliveries a year.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
preeclampsia | From date of randomization until the date of delivery

SECONDARY OUTCOMES:
birth weight | at delivery, assessed up to 40 weeks
preterm birth | at delivery, assessed up to 40 weeks
gestational diabetes | From date of randomization until the date of delivery

CONTACTS AND LOCATIONS:
Overall Officials: yves jacquemyn, PhD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

REFERENCES:
- [Derived] Verheyen VJ, Remy S, Lambrechts N, Govarts E, Colles A, Poelmans L, Verachtert E, Lefebvre W, Monsieurs P, Vanpoucke C, Nielsen F, Van den Eeden L, Jacquemyn Y, Schoeters G. Residential exposure to air pollution and access to neighborhood greenspace in relation to hair cortisol concentrations during the second and third trimester of pregnancy. Environ Health. 2021 Feb 11;20(1):11. doi: 10.1186/s12940-021-00697-z. PMID 33573648